CLINICAL TRIAL: NCT05154591
Title: Chronic Kidney Disease of Unknown Cause (CKDu) Treated With Directed Local Intra-arterial Infusion of Autologous Stromal Vascular Fraction (SVF) Cells.
Brief Title: CKDu Treated With Intra-arterial Infusion of Autologous SVF Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samuel Vilchez, PhD (Other)
Collaborators: Ministerio de Salud de Nicaragua (Unknown); GID BIO (Unknown); National Autonomous University of Nicaragua (Other)
Responsible Party: Sponsor-Investigator, Samuel Vilchez, PhD, Professor, National Autonomous University of Nicaragua
Organization: National Autonomous University of Nicaragua (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVF2015MeN-1
Record Dates: First submitted 2021-11-06; First posted 2021-12-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Chronic Renal Failure of Unknown Cause
Keywords: Stromal vascular fraction; Mesenchynmal stem cells; Chronic kidney disease; Adipose stem cells
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Masking Description: * Open label for surgeons and radiologists
  * Closed label for pathologists and nephrologists
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral Treatment (Experimental): Intra-arterial injection of SVF cells into the kidneys.
  Interventions: Genetic: Adipose-derived stromal vascular fraction cells

INTERVENTIONS:
Genetic: Adipose-derived stromal vascular fraction cells — Kidney structural and functional changes in 18 patients after 36 months of treatment with SVF cells.

SUMMARY:
This is an interventional study to treat 18 patients with chronic kidney disease of unknown cause (CKDu), formerly known as Mesoamerican nephropathy (MeN), with autologous adipose tissue-derived stromal vascular fraction (SVF) cells transplanted by intra-arterial injection both kidneys.

This study assesses: (1) safety and tolerability, (2) preliminary evidence of efficacy, (3) exploratory evidence of clinical effects.

DETAILED DESCRIPTION:
Patients under go 24 hours of preoperative hydration combined with N-actyl cysteine 300 mg IV for prevention of nephrotoxicity. Under general anesthesia 200-300 cc of lipoaspirate is collected into a sterile processing cannister (GID SFV-1, Louisville, CO, USA). The tissue is washed and dissociated with collagenase (Worthington CLS-1, Lakewood, NJ, USA) at a concentration of 200 CDU/ml of total volume for 50 minutes at 39°C. This is followed by inactivation using 40 cc of human serum albumin. SVF cells are separated via centrifugation for 10 minutes at 800 g. The cell pellet is extracted and resuspended in Harmann solution with an aliquot (10 µl) removed for counting and viability assessment of resulting total nucleated cells (YNC) through and image cytometer (ADAM MC, Portsmouth NH, USA).

Femoral artery catheterization is performed permitting advancement of a 100 cc balloon-tip catheter into the renal artery under fluoroscopic control, with position confirmation using 1 cc of OrtoRay® 320 contrast diluted 1:4 with Hartmann solution. SVF cells are then admixed with 200 cc Hartmann solution warmed to 37°C and in fused using a DRE infusion pump (DRE Medical, Louisville, KY, USA) over a 15 minute period with constant agitation. On the 1st pos-operative day creatinine and glomerular filtration rate are checked and the patient is discharged.

Follow-up studies include clinical assessment, chemistries, and renal ultrasound to assess intra-parenchymal renal volume, renal blood flow distribution, and hilar artery vascular resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mesoamerican nephropathy
* Stages 3 and 4
* No other renal disease
* No essential hypertension

Exclusion Criteria:

* Significant abnormalities in laboratory tests that contraindicate surgical procedures.
* Acute pathology or complications of significant chronic pathologies in the 6 months prior to study entry, including, but not limited to:

Medical history of deep vein thrombosis Uncontrolled hypertension Active infection Reduced cardiac ejection fraction Hepatitis B, C or HIV Diabetes treated with insulin or glucose lowering agents Anemia (Hb <9 g/dL) History of cancer Severe depression (Beck scale) Autoimmune disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | 36-months follow-up post intervention.
  Documentation of adverse events
Preliminary evidence of efficacy | Assessment of changes between day 7 and month 36 post intervention.
  Improvement in clinical parameter of GFR as compared with historical age and stage-matched controls.

SECONDARY OUTCOMES:
Renal blood flow. | Up to month 12 post intervention.
  Distribution of intra-renal blood flow.
Kidney volume. | Up to month 12 post intervention.
  Changes in kidney size (cm3).
Renal arterial resistive index. | Up to month 12 post intervention.
  Decreases in hilar artery resistance index (less o equal to 0.7).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Carstens, MD, Principal Investigator — Wake Forrest Institute for Regenerative Medicine; Diego Correa, MD, PhD, Principal Investigator — University of Miami; Sreedhar Mandayam, MD, Study Director — University of Texas
Locations (1):
- Hospital Escuela Oscar Danilo Rosales Arguello, León, Nicaragua

REFERENCES:
- [Result] Brown JC, Shang H, Li Y, Yang N, Patel N, Katz AJ. Isolation of Adipose-Derived Stromal Vascular Fraction Cells Using a Novel Point-of-Care Device: Cell Characterization and Review of the Literature. Tissue Eng Part C Methods. 2017 Mar;23(3):125-135. doi: 10.1089/ten.TEC.2016.0377. PMID 28177263
- [Result] Caplan AI, Correa D. The MSC: an injury drugstore. Cell Stem Cell. 2011 Jul 8;9(1):11-5. doi: 10.1016/j.stem.2011.06.008. PMID 21726829
- [Result] Carstens MH, Quintana FJ, Calderwood ST, Sevilla JP, Rios AB, Rivera CM, Calero DW, Zelaya ML, Garcia N, Bertram KA, Rigdon J, Dos-Anjos S, Correa D. Treatment of chronic diabetic foot ulcers with adipose-derived stromal vascular fraction cell injections: Safety and evidence of efficacy at 1 year. Stem Cells Transl Med. 2021 Aug;10(8):1138-1147. doi: 10.1002/sctm.20-0497. Epub 2021 Apr 7. PMID 33826245
- [Result] Correa-Rotter R, Garcia-Trabanino R. Mesoamerican Nephropathy. Semin Nephrol. 2019 May;39(3):263-271. doi: 10.1016/j.semnephrol.2019.02.004. PMID 31054625
- [Result] Guo J, Nguyen A, Banyard DA, Fadavi D, Toranto JD, Wirth GA, Paydar KZ, Evans GR, Widgerow AD. Stromal vascular fraction: A regenerative reality? Part 2: Mechanisms of regenerative action. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):180-8. doi: 10.1016/j.bjps.2015.10.014. Epub 2015 Oct 24. PMID 26546112
- [Result] Johnson RJ, Wesseling C, Newman LS. Chronic Kidney Disease of Unknown Cause in Agricultural Communities. N Engl J Med. 2019 May 9;380(19):1843-1852. doi: 10.1056/NEJMra1813869. No abstract available. PMID 31067373
- [Result] Nguyen A, Guo J, Banyard DA, Fadavi D, Toranto JD, Wirth GA, Paydar KZ, Evans GR, Widgerow AD. Stromal vascular fraction: A regenerative reality? Part 1: Current concepts and review of the literature. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):170-9. doi: 10.1016/j.bjps.2015.10.015. Epub 2015 Oct 31. PMID 26565755
- [Result] Wijkstrom J, Gonzalez-Quiroz M, Hernandez M, Trujillo Z, Hultenby K, Ring A, Soderberg M, Aragon A, Elinder CG, Wernerson A. Renal Morphology, Clinical Findings, and Progression Rate in Mesoamerican Nephropathy. Am J Kidney Dis. 2017 May;69(5):626-636. doi: 10.1053/j.ajkd.2016.10.036. Epub 2017 Jan 23. PMID 28126239